CLINICAL TRIAL: NCT06985212
Title: Study of the Natural History of Acid Sphingomyelinase Deficiency (ASMD): National, Multicenter Cohort of Adult and Pediatric Patients _FASMD (French Prospective Cohort ASMD)
Brief Title: National Multicentre Study of the Natural History of Acid Sphingo-myelinase Deficiency in Adults and Children
Acronym: FASMD
Status: Not yet recruiting | Type: Observational
Sponsor: Wladimir MAUHIN, Dr (Other)
Collaborators: Beaujon Hospital (Other); University Hospital, Montpellier (Other); Centre Hospitalier Saint Joseph Saint Luc de Lyon (Other); Bichat Hospital (Other); Versailles Hospital (Other); University Hospital, Bordeaux (Other); Hôpital de la Timone (MARSEILLE) (Unknown); Hôpital Claude-Huriez (Other); Hospices Civils de Lyon (Other); Hôpital Armand Trousseau (Other); Centre Hospitalier de Cornouaille (Other); Nantes University Hospital (Other); University Hospital, Angers (Other Government); Hospital BLOIS (Unknown); Hôpital Pasteur, CHU Nice (Unknown); Centre Hospitalier Eure-Seine (Other); University Hospital, Orléans (Unknown); University Hospital, Toulouse (Other); APHM - Nord (Unknown); Henri Mondor University Hospital (Other); Hôpital Européen Marseille (Other); CH Henri Mondor (Aurillac) (Unknown); University Hospital, Clermont-Ferrand (Other); Centre Hospitalier Universitaire de Saint Etienne (Other); Hôpital Pellegrin, CHU Bordeau (Unknown); Reims University hospital (Other); Hospital Avicenne (Other); University Hospital, Strasbourg (Other); Necker Hospital, 75015 Paris (Unknown)
Responsible Party: Sponsor-Investigator, Wladimir MAUHIN, Dr, Principal Investigator, Groupe Hospitalier Diaconesses Croix Saint-Simon
Organization: Groupe Hospitalier Diaconesses Croix Saint-Simon (Other)
Other Study IDs: 2024-A01376-41
Record Dates: First submitted 2025-03-18; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-03

CONDITIONS: Acid Sphingomyelinase Deficiency (ASMD); Niemann Pick Disease
Keywords: ASMD; ASMD Pick A/A-B/B; registry; database
MeSH Terms: conditions — Niemann-Pick Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 120 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Experimental Cohort: A cohort of 200 pediatric and adult participants, diagnosed of ASMD, as established by a confirmed low acid sphingomyelinase assay, and who have not given their opposition (patient and/or parent) to participate in this research.

SUMMARY:
The goal of this study is to describe the natural history of ASMD in adult and paediatric patients with or without specific treatment in order to assess the impact of the disease on their daily lives and quality of life.

The population concerned corresponds to patients aged at least 2 years, with a definite diagnosis of ASMD as determined by a confirmed low acid sphingomyelinase assay and who have not expressed their opposition to participating in this research (patients and/or parental authority).

DETAILED DESCRIPTION:
Niemann Pick A/ AB/ B disease also known as acid sphingomyelinase deficiency (ASMD) is a very rare genetic disease. The natural history remains poorly understood. This disease leads to morbidity and mortality. A specific effective treatment has been available since 2023.

The Internal Medicine Department of the Groupe Hospitalier Diaconesses Croix Saint-Simon (GHDCSS), reference center for lysosomal diseases, develops this clinical study in order to better understand the natural history of Niemann Pick A/ AB/ B disease, and better manage the symptoms, the complications and also the impact of this new treatment, particularly on daily life (quality of life). This French multicenter cohort research is coordinated by Dr Wladimir MAUHIN, (Internal medicine department, GHDCSS, Paris).

ELIGIBILITY:
Inclusion Criteria:

1. Any patient aged at least 2 years, with a confirmed diagnosis of ASMD determined by a lowered acid sphingomyelinase assay.
2. Have received written and oral information about the protocol and have not expressed opposition to participating in the study.
3. Affiliated to the social security system or entitled to benefits (excluding AME).

Exclusion Criteria:

1. Inability to understand the information provided,
2. Under guardianship, trusteeship or judicial protection,
3. Under detention or deprived of liberty by judicial or administrative decision.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population will be patients aged 2 years or older with a definite diagnosis of ASMD, as determined by a confirmed low acid sphingomyelinase assay, and who have not given their opposition (patient and/or parent) to participate in this research.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2035-04-15 (Estimated); Study Completion 2035-04-15 (Estimated)

PRIMARY OUTCOMES:
To describe the natural history of ASMD (symptoms, complications) | 120 months
  To describe the natural history of ASMD (symptoms, complications) in adult and paediatric patients with and without therapeutic treatment and to assess their quality of life.

SECONDARY OUTCOMES:
Identify of prognostic factors, available treatments and phenotypic forms of the disease | 120 months
  * Identify prognostic factors for the disease: genetic, biochemical, symptomatic, radiological and social.
  * Evaluate the therapeutic treatments available.
  * List the different phenotypic forms on a national scale.
  * To highlight the social problems associated with the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Wladimir Mauhin, MD PhD, Study Director — Groupe Hospitalier Diaconesses Croix Saint-Simon
Locations (1):
- Groupe Hospitalier Diaconesses Croix Saint-Simon, Paris, France, France

IPD SHARING:
Plan to Share IPD: Undecided
undefined